CLINICAL TRIAL: NCT01532635
Title: A Two Step Approach to Allogeneic Hematopoietic Stem Cell Transplantation for High-Risk Hematologic Malignancies Using Two Related Donors
Brief Title: A Two-Step Approach to Bone Marrow Transplant Using Cells From Two Partially-Matched Relatives
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11D.570; 2011-101 (Other: CCRRC); JT 1832 (Other: JeffTrial Number)
Record Dates: First submitted 2012-02-06; First posted 2012-02-14 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Malignancy; Leukemia; Acute Lymphoblastic Leukemia; ALL; Acute Myelogenous Leukemia; AML; Chronic Lymphocytic Leukemia; CLL; Lymphoma; Hodgkin's Lymphoma; Non-hodgkin's Lymphoma; Myeloma
Keywords: hematologic malignancy; leukemia; Acute lymphoblastic leukemia; ALL; Acute myelogenous leukemia; AML; Chronic lymphocytic leukemia; CLL; lymphoma; hodgkin's lymphoma; non-hodgkin's lymphoma; myeloma; allogeneic stem cell transplant; TJU 2-step; Hematopoietic stem cell transplant; HSCT; bone marrow transplant; Cyclophosphamide; MMF; Mycophenolate Mofetil
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell | interventions — Whole-Body Irradiation; Radiotherapy; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic HSCT Using Two Related Donors (Experimental): CONDITIONING: Patients undergo TBI BID on days -9 to -6, undergo DLI on day -6, and receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANTATION: Patients undergo CD34+ selected allogeneic HSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO beginning on day -1 with taper beginning on day 42 and mycophenolate mofetil IV or PO BID on days -1 to 28.
  Interventions: Radiation: Total Body Irradiation (TBI); Biological: Donor Lymphocyte Infusion (DLI); Drug: Cyclophosphamide (CY); Drug: Tacrolimus; Drug: Mycophenolate Mofetil (MMF); Biological: Hematopoietic Stem Cell Transplant (HSCT)

INTERVENTIONS:
Radiation: Total Body Irradiation (TBI) — TBI twice daily for 4 days and occurs 6 to 9 days prior to the transplant. Total radiation dose is 12 Gy.
  Other Names: TBI; radiotherapy
Biological: Donor Lymphocyte Infusion (DLI) — DLI given 6 days prior to transplant (HSCT).
  Other Names: DLI; T cell infusion
Drug: Cyclophosphamide (CY) — Cyclophosphamide given once daily at 60 mg/kg on days 2 and 3 prior to transplant (HSCT).
  Other Names: CY; Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Tacrolimus — Tacrolimus is started the day before the transplant and stops a few months after transplant.
  Other Names: FK-506; fujimycin; Prograf; Advagraf; Protopic
Drug: Mycophenolate Mofetil (MMF) — MMF is started the day before transplant and stops a few weeks after transplant.
  Other Names: MMF; CellCept; Myfortic
Biological: Hematopoietic Stem Cell Transplant (HSCT) — CD34+ selected Hematopoietic Stem Cell Transplant (HSCT) is performed using donor cells from two related donors.
  The CliniMACS® Plus Instrument will be used for the selection of human CD34+ hematopoietic stem cells.
  Other Names: HSCT; stem cell transplant; CliniMACS

SUMMARY:
This phase II clinical trial studies how well two donors stem cell transplant work in treating patients with high-risk hematologic malignancies. After receiving radiation to help further treat the disease, patients receive a dose of donors' T cells. T cells can fight infection and react against cancer cells. Two days after donors' T cells are given, patients receive cyclophosphamide (CY) to help destroy the most active T cells that may cause tissue damage (called graft versus host disease or GVHD). Some of the less reactive T cells are not destroyed by CY and they remain in the patient to help fight infection. A few days after the CY is given, patients receive donors' stem cells to help their blood counts recover. Using two donors' stem cell transplant instead of one donor may be more effective in treating patients with high-risk disease and may prevent the disease from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess 1 year relapse free survival in patients undergoing hematopoietic stem cell transplant (HSCT) using the Thomas Jefferson University (TJU) 2 step approach using 2 donors.

SECONDARY OBJECTIVES:

I. To assess the consistency and pace of engraftment. II. To assess the pace of T cell and B cell immune recovery in patients in each arm.

III. To assess regimen related toxicity, graft-versus-host disease (GVHD) incidence and severity, and overall survival.

IV. To assess the tolerance of the period of fever, diarrhea, and rash after the introduction of second donor and qualitatively compare it to prior patient groups or concurrent patient groups.

V. To assess chimerism to ascertain whether one donor is emerging as dominant at regular intervals beginning at the time of engraftment.

VI. If dominance is observed, to compare the donors with regard to degree of human leukocyte antigen (HLA) mismatch, killer Ig-like receptor (KIR) types, cluster of differentiation (CD)34+ cell doses, infusion order, donor age, and donor alloreactivity points in an effort to identify potential biologic factors that predict for dominance. To determine if trends toward dominance occur in T cell, natural killer (NK) cell, or other cellular subsets prior to emerging in the graft as a whole.

VII. To assess if establishment of a dominant donor versus persistent chimerism of both donors is associated with a lower relapse rate.

VIII. To collect leukemia samples prior to transplant and after relapse whenever possible. To assess the overall degree of HLA-class I and class II expression on these paired samples. To test for loss of one or both HLA haplotypes in the relapsed tumor specimens. When observed, to correlate loss of one HLA haplotype with: a) receipt of a transplant capable of targeting only that haplotype; b) establishment of dominance in a 2 haplotype transplant such that the lost haplotype would be the primary target of the dominant donor; c) being the target of the donor predicted to be more alloreactive in a 2 haplotype transplant.

OUTLINE:

CONDITIONING: Patients undergo total-body irradiation (TBI) twice daily (BID) on days -9 to -6, undergo donor lymphocyte infusion (DLI) on day -6, and receive cyclophosphamide intravenously (IV) over 2 hours on days -3 and -2.

TRANSPLANTATION: Patients undergo CD34+ selected allogeneic HSCT on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV or orally (PO) beginning on day -1 with taper beginning on day 42 and mycophenolate mofetil IV or PO BID on days -1 to 28.

After completion of study treatment, patients are followed up for 1 year, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematologic malignancy with residual disease (morphological, cytogenetic, molecular, or radiographic) after treatment with 1 or more chemotherapy regimens in whom achievement of remission with additional chemoradiotherapy is felt to be unlikely or who is in 3rd or greater CR. Patients with marrow based diseases in which the marrow biopsy does not meet criteria for active disease (i.e. <5% blasts in acute leukemia) but who does not have full count recovery will be eligible for treatment on this high risk trial.
2. Patients must have two related donors that meet an acceptable scenario as described above.
3. Patients must adequate organ function:

   * LVEF of >= 50%
   * DLCO (adjusted for hemoglobin) >= 50% of predicted
   * Adequate liver function as defined by a serum bilirubin =< 1.8, AST or ALT < 2.5X upper limit of normal
   * Creatinine clearance of >= 60 ml/min
4. Karnofsky Performance Status of > 80 % on the modified KPS tool (see Appendix A).
5. Patients must be willing to use contraception if they have childbearing potential.
6. Able to give informed consent

Exclusion Criteria:

1. Modified KPS of < 80%
2. >= 5 Comorbidity Points on the HCT-CI Index (See Appendix B)
3. Class I or II antibodies against donor HLA antigens
4. HIV positive
5. Active involvement of the central nervous system with malignancy
6. Psychiatric disorder that would preclude patients from signing an informed consent
7. Pregnancy, or unwillingness to use contraception if they have child bearing potential
8. Patients with life expectancy of =< 6 months for reasons other than their underlying hematologic/oncologic disorder
9. Alemtuzumab treatment within 8 weeks of HSCT admission.
10. ATG level of >= 2 ugm/ml
11. Patients with active inflammatory processes (such as flair of an autoimmune disease) including T max > 101, or active tissue inflammation are excluded.
12. Inability to tolerate cyclophosphamide or undergo total body irradiation at the doses specified in the treatment plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University; Dolores Grosso, DNP, CRNP, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogeneic HSCT Using Two Related Donors
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.35 (20.64)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: One Year Relapse-Free Survival
Description: To assess one year relapse-free survival (RFS) in patients undergoing HSCT (hematopoietic stem cell transplantation) using the TJU 2 step-approach with two donors.
  Survival will be estimated by the Kaplan-Meier method. All estimates of rates will be presented with corresponding confidence intervals. For 1 year RFS rates, the method of Atkinson and Brown will be used to allow for the two-stage design; otherwise the method of Conover.
Time Frame: 1 year
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

2. Secondary Outcome: Chimerism Assessment
Description: To assess chimerism to ascertain whether one donor is emerging as dominant at regular intervals beginning at the time of engraftment.
Time Frame: 1 year
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

3. Secondary Outcome: Assessment of Dominance
Description: If dominance is observed, to compare the 2 donors with regard to degree of HLA mismatch, KIR types, CD 34+ cell doses, infusion order, donor age, and donor alloreactivity points in an effort to identify potential biologic factors that predict for dominance. To determine if trends toward dominance occur in T cell, NK cell, or other cellular subsets prior to emerging in the graft as a whole.
Time Frame: 1 year
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

4. Secondary Outcome: Relapse Rates
Description: To assess if establishment of a dominant donor versus persistent chimerism of both donors is associated with a lower relapse rate.
Time Frame: 1 year
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

5. Secondary Outcome: Engraftment
Description: To assess the consistency and pace of engraftment of both donors.
Time Frame: 1 year
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

6. Secondary Outcome: Immune Reconstitution
Description: Assess T and B cell Reconstitution
Time Frame: 1 year
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

7. Secondary Outcome: Non-relapse Morbidity and Mortality
Description: Assessment of regimen related toxicity, GVHD incidence and severity, and overall survival.
Time Frame: 1 year
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

8. Secondary Outcome: Tolerance of DLI
Description: Assessment of the tolerance of the period of fever, diarrhea, and rash after the introduction of second donor and qualitatively compare it to prior patient groups or concurrent patient groups
Time Frame: 2-6 days prior to transplant
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

9. Secondary Outcome: Assessment for Tumor Escape Mechanisms
Description: To test for loss of one or both HLA haplotypes in patients who relapse post-transplant and examine the relapse in the context of the characteristics of the 2 donors
Time Frame: 1 year post transplant
Arm/Group | Allogeneic HSCT Using Two Related Donors
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Allogeneic HSCT Using Two Related Donors
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic HSCT Using Two Related Donors (N=4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fevers (General disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Blood and lymphatic system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic HSCT Using Two Related Donors (N=4)
Abdominal pain (General disorders) | 2 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Arm pain (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (General disorders) | 2 (2)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Balance problems (General disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Change in vision (Eye disorders) | 1 (1)
Chest pain (General disorders) | 3 (4)
Chest tightness (General disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Clostridium difficile (Gastrointestinal disorders) | 1 (1)
CMV reactivation (Immune system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (4)
Decreased urine output (Renal and urinary disorders) | 2 (4)
Dehydration (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (9)
Dizziness (General disorders) | 1 (1)
Dry eyes (General disorders) | 1 (1)
Dyspepsea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (4)
Edema (Skin and subcutaneous tissue disorders) | 1 (1)
Electrolyte imbalance (Blood and lymphatic system disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Feet pain (General disorders) | 1 (1)
Fevers (General disorders) | 4 (11)
Fluid overload (Blood and lymphatic system disorders) | 2 (3)
Generalized pain (General disorders) | 2 (2)
Generalized weakness (General disorders) | 1 (1)
GVHD rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hand pain (General disorders) | 1 (1)
Headache (General disorders) | 3 (3)
Heartburn (Gastrointestinal disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
HHV-6 reactivation (Blood and lymphatic system disorders) | 1 (1)
Hiccups (General disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 4 (6)
Hypertension (Blood and lymphatic system disorders) | 2 (3)
Hypokalemia (Blood and lymphatic system disorders) | 1 (2)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 3 (5)
Hypothermia (General disorders) | 1 (1)
Hypoxia (Blood and lymphatic system disorders) | 2 (3)
Increased alkaline phosphatase (General disorders) | 1 (1)
Increased creatinine (Blood and lymphatic system disorders) | 3 (4)
Increased LFTs (Hepatobiliary disorders) | 1 (1)
Knee pain (General disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 4 (4)
Neck pain (General disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2)
Orthostatic hypotension (Blood and lymphatic system disorders) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Parotitis (General disorders) | 1 (1)
Platelet transfusion reaction (Blood and lymphatic system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (9)
Rectal pain (General disorders) | 1 (1)
Rigors (General disorders) | 1 (1)
Shoulder pain (General disorders) | 1 (1)
Swollen ankles (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Toenail bleeding (General disorders) | 1 (1)
Trouble sleeping (General disorders) | 2 (2)
Upper extremity swelling (General disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Vaginal discomfort/itching (General disorders) | 1 (1)
Volume overload (Cardiac disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to poor accrual. No reportable data has been collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes